CLINICAL TRIAL: NCT01225341
Title: A Double-Blind, Randomized, Placebo Controlled, Crossover Study to Assess the Safety and Efficacy of Botulinum Toxin A Injections as a Preventative Measure for Herpes Labialis.
Brief Title: Botulinum Toxin A for Herpes Labialis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too many patients withdrew/lost to follow up
Sponsor: DeNova Research (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HSV-BOT-01-09
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Herpes Labialis
Keywords: HSV-1; Herpes labialis; Cold sores; Fever blisters
MeSH Terms: conditions — Herpes Labialis | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- onabotulinumtoxinA/placebo (Experimental): Patients will be injected every 3 months with onabotulinumtoxinA for a period of 12 months. At the 12 month visit, patients will receive injections of saline.
  Interventions: Drug: onabotulinumtoxinA; Other: Bacteriostatic normal saline
- Bacteriostatic normal saline/ onabotulnimtoxinA (Placebo Comparator): Patients will be injected every 3 months with saline for a period of 12 months. At the 12 month visit, patients will receive injections of onabotulnimtoxinA.
  Interventions: Drug: onabotulinumtoxinA; Other: Bacteriostatic normal saline

INTERVENTIONS:
Drug: onabotulinumtoxinA — Botox® is supplied in a 100 U vial and will be reconstituted with 3.3 mL of 0.9% Sodium Chloride Injection USP to yield a solution of 3 U per 0.1 mL. Study treatment will consist of an injection of Botox® (onabotulinumtoxinA) (3 U/ 0.1 mL) into the orbicularis oris muscle (8 U, .27 mL in the upper and/or lower lip, depending on the site of recurrence) using a 30G needle.
  Other Names: Botox
Other: Bacteriostatic normal saline — Study treatment will consist of an injection of bacteriostatic normal saline, into the orbicularis oris muscle (8 U, .27 mL in the upper and/or lower lip, depending on the site of recurrence) using a 30G needle.
  Other Names: Saline

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Botulinum Toxin Type A as a preventative measure for Herpes Labialis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 64.
* Have herpes simplex virus 1 (HSV-1) with between 2-6 herpes labialis recurrences per year.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following is documented on the medical history:
* postmenopausal for at least 12 months prior to study drug administration
* without a uterus and/or both ovaries
* has had a bilateral tubal ligation for at least 6 months prior to study drug administration.
* absence of an other physical condition according to the PI's discretion
* Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

* Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
* Subjects with a known allergy or sensitivity to any component of the study medications or anesthesia.
* Active recurrence of herpes labialis.
* Botulinum toxin to the lower 1/3 of the face with the past 6 months.
* Significant concurrent illness such as diabetes, epilepsy, lupus, or congestive heart failure.
* Concurrent skin condition affecting area to be treated.
* Prior surgery on the area to be treated within 3 months of initial treatment or during the study.
* History or evidence of keloids or hypertrophic scarring.
* Current use of antivirals for the treatment of herpes labialis within 2 weeks prior to initiation of treatment (e.g., acyclovir, valaciclovir, famciclovir, and penciclovir).
* Topical use of over-the-counter medications for the treatment or prevention of HSV-1 (e.g., Abreva).
* Subjects currently using aminoglycoside antibiotics, curare-like agents or other agents that might interfere with neuromuscular function.
* Subjects with a diagnosis of Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function or current facial palsy.
* Current history of chronic drug or alcohol abuse.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Subjects who, in the Investigator's opinion, have a history of poor cooperation, non-compliance with medical treatment or unreliability.
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research/ Chicago Center for Facial Plastic Surgery
Locations (1):
- DeNova Research, Chicago, Illinois, United States

REFERENCES:
- See also: DeNova Research — http://www.denovaresearch.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Period: Overall Study
Arm/Group | onabotulinumtoxinA/Placebo | Bacteriostatic Normal Saline/ onabotulnimtoxinA
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA/Placebo | Bacteriostatic Normal Saline/ onabotulnimtoxinA | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — Population: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Age, Continuous — Population: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Sex: Female, Male — Population: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Region of Enrollment [unit: participants] — Population: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Recurrence and Duration of Herpes Labialis Lesions
Description: Days between last injection and outbreak onset & Days between onset and recurrence
Time Frame: 12 months
Population: as for baseline characteristics
Groups:
- OnabotulinumtoxinA: Patients will be injected every 3 months with onabotulinumtoxinA for a period of 12 months.
  OnabotulinumtoxinA: Botox® is supplied in a 100 U vial and will be reconstituted with 3.3 mL of 0.9% Sodium Chloride Injection USP to yield a solution of 3 U per 0.1 mL. Study treatment will consist of an injection of Botox® (onabotulinumtoxinA) (3 U/ 0.1 mL) into the orbicularis oris muscle (8 U, .27 mL in the upper and/or lower lip, depending on the site of recurrence) using a 30G needle.
- Bacteriostatic Normal Saline: Patients will be injected every 3 months with saline for a period of 12 months.
  Bacteriostatic normal saline: Study treatment will consist of an injection of bacteriostatic normal saline, into the orbicularis oris muscle (8 U, .27 mL in the upper and/or lower lip, depending on the site of recurrence) using a 30G needle.
Arm/Group | OnabotulinumtoxinA | Bacteriostatic Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Measurement of Lesion Size
Description: Lesions will be measured in millimeters across the maximal lesion length in mm
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | OnabotulinumtoxinA | Bacteriostatic Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pain Assessment
Description: Each day of a recurrence of herpes labialis, the subject will document his/her pain level in the diary according to the Visual Analog Scale for pain (VAS) by placing a straight line intersecting the pain line. The scale will be 10 cm long and the distance from start to mark will be measured in millimeters.
  Score range is 0-10. Scores closer to 0 signify lower pain levels and scores closer to 10 signify high pain levels
Time Frame: During outbreak
Population: as for baseline characteristics
Arm/Group | OnabotulinumtoxinA | Bacteriostatic Normal Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Symptom Evaluation
Description: Each day of a recurrence of herpes labialis, the subject will document his/her pain level in the diary according to a 4-point scale ((0) none, (1) mild, (2) moderate, (3) severe).
  Scores closer to 0 indicate a more favorable outcome.
Time Frame: During outbreak
Population: as for baseline characteristics
Arm/Group | OnabotulinumtoxinA | Bacteriostatic Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Description: The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report
Arm/Group | onabotulinumtoxinA | Bacteriostatic Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated and the PI/study team no longer has access to study data as it was destroyed. Efforts were exhausted to locate any remaining data, but were unsuccessful. No study data are available to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes